CLINICAL TRIAL: NCT04452851
Title: Portable Non-invasive Positive Pressure Airway Device Therapy System Efficacy Study
Brief Title: Portable Positive Pressure Therapy Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koronis Biomedical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: R44HL154932 (NIH)
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Subjects will be asked to participate in four (4) visits. During the first visit, baseline measurements will be made. In the subsequent three (3) sessions, subjects will be asked to perform two (2) tests from a group of six (6) options. This list of tests is comprised of three BiPAP Equivalency tests and three Activity of Daily Living Simulations. Participants will be randomized to study groups using a table of random numbers generated at the outset of the study to determine the test order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (6):
- Treadmill test with BREATHE (Experimental): Subjects will perform exercise tests identical to the treadmill tests from the baseline test. However, in this test, after they reach a Borg score of 7, they will be allowed to recover with the prototype BREATHE system until they are fully recovered (Borg: 0).
  Interventions: Device: BREATHE
- Treadmill test with BiPAP (Active Comparator): Subjects will perform exercise tests identical to the treadmill tests from the baseline test. However, in this test, after they reach a Borg score of 7, they will be allowed to recover with a standard BiPAP machine until they are fully recovered (Borg: 0).
  Interventions: Device: BiPAP
- Treadmill test with placebo inhaler (Placebo Comparator): Subjects will perform exercise tests identical to the treadmill tests from the baseline test. However, in this test, after they reach a Borg score of 7, they will be allowed to recover with a placebo inhaler until they are fully recovered (Borg: 0).
  Interventions: Drug: COPD Inhaler
- Activity of Daily Living with BREATHE (Experimental): Subjects will be asked to complete Glittre-ADL tests with the BREATHE system being available for use throughout the test and recovery period. Borg scores will be measured after each minute of exercise and every 30 seconds during seated recovery until the subject is fully recovered (Borg: 0).
  Interventions: Device: BREATHE
- Activity of Daily Living with BREATHE during recovery (Experimental): Subjects will be asked to complete Glittre-ADL tests with the BREATHE system being available for use throughout the test and recovery period. Borg scores will be measured after each minute of exercise and every 30 seconds during seated recovery until the subject is fully recovered (Borg: 0).
  Interventions: Device: BREATHE
- Activity of Daily Living (No Intervention): Subjects will be asked to complete Glittre-ADL tests with the BREATHE system will NOT be available for use throughout the test and recovery period. Borg scores will be measured after each minute of exercise and every 30 seconds during seated recovery until the subject is fully recovered (Borg: 0).

INTERVENTIONS:
Device: BREATHE — The on-demand handheld portable noninvasive positive pressure airway device unit generates BiPAP by using a built-in blower which intakes air from the nearby ambient. The BiPAP pressure functions as a virtual stent within the lungs of a user with COPD. The virtual stent opens the passageways within the user lungs. Once opened, the virtual stent facilitates gas exchange in order to relieve dyspnea. By temporarily facilitating this gas exchange, the user will quickly recover from dyspnea in order to resume regular activities.
  Arms: Activity of Daily Living with BREATHE; Activity of Daily Living with BREATHE during recovery; Treadmill test with BREATHE
Device: BiPAP — BiPAP stands for Bilevel Positive Airway Pressure, and is very similar in function and design to a CPAP machine (continuous positive airway pressure). A BiPAP machine is a non-invasive form of therapy for patients suffering from sleep apnea.
  Arms: Treadmill test with BiPAP
Drug: COPD Inhaler — Inhaler medication to support quick relief from COPD symptoms
  Arms: Treadmill test with placebo inhaler

SUMMARY:
This study will assess the impact the BREATHE device provides on post-exertion recovery time in COPD patients when used during and/or after performing an Activity of Daily Living simulation. It will also establish equivalency with BiPAP machines.

DETAILED DESCRIPTION:
Study Overview: Potential subjects who are clinically stable COPD patients with 30% ≤ FEV1 < 50% (COPD GOLD criteria stage 3), will be enrolled. Following consent procedures, interested participants will be screened for eligibility. Eligible subjects will be invited to the test facility for four (4) visits. During the first visit, baseline measurements will be made. In the subsequent three (3) sessions, subjects will be asked to perform two (2) tests (BiPAP Equivalency Test and Activity of Daily Living Simulation). Baseline evaluation techniques will include spirometry, a Six Minute Walk Test (6MWT) (which produces a Six Minute Walk Distance, or 6MWD), and finally, a baseline treadmill test. Prior to the baseline treadmill test, Borg Scores will be measured. The subjects will then be asked to walk at a comfortable speed on the treadmill. The incline will be increased each minute by either 1% (Baseline 6MWD < 250m) or 2% (Baseline 6MWD >250m) until they reached a Borg score of 7.

In subsequent visits, subjects will be randomly assigned each of six tests including: treadmill tests that repeat the baseline treadmill test with a) the prototype BREATHE device, b) a standard BiPAP system, or c) a placebo inhaler used during recovery; and Glittre ADL tests where the subject either has access to the BREATHE device a) withheld, b) during recovery, and c) during test performance and recovery. The primary endpoint in each of these tests is the recovery time (return to 0 Borg, "No difficulty breathing"). SpO2, heart rate, respiration rate, and total test times will also be recorded during each test.

BiPAP Equivalency Test: Subjects will perform exercise tests identical to the treadmill tests from the baseline test. However, in these tests, after they reach a Borg score of 7, they will be allowed to recover with a) the prototype BREATHE system, b) a standard BiPAP machine, and c) a placebo inhaler until they are fully recovered (Borg: 0).

Activity of Daily Living Simulation: Subjects will be asked to complete Glittre-ADL tests. This test is a standard COPD functional performance instrument. At the beginning of each test, participants will be instructed to rise from a chair and walk 10 meters, ascending a 2-step rise about half-way along that distance, to reach a shelving unit. The shelves will be positioned at shoulder and waist height. The participant will move 3 cartons, each weighing 1 kg, from the upper to the lower shelf and then to the floor.

The sequence is then reversed so that each carton is returned to the top shelf before the participant returns to the starting position at the chair. At that time the participant sits down and then immediately rises to begin the next lap. The test ends when the participant completes 5 of these laps. Participants are told to perform the test as quickly as possible. Rests are allowed but participants are told to resume activity as soon as possible. During the test, participants will wear a backpack filled with a 2.5 (women) or 5 kg (men) weight. The 2.5 kg weight simulates the weight of a supplemental oxygen unit, which can be exchanged for the weight when appropriate. This allows the addition of oxygen for future tests without affecting the integrity of the test.

Three different Glittre-ADL tests will be completed. In these sessions, the BREATHE system will a) not be available, b) be available for use during post-exertion recovery, and c) be available for use throughout the test and recovery period. Borg scores will be measured after each minute of exercise and every 30 seconds during seated recovery until the subject is fully recovered (Borg: 0).

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 21 to 85
* Clinically stable
* Diagnosis of COPD following ERS-ATS guidelines 2011 update with GOLD criteria stage 3 ("Severe"), 30% ≤ FEV1 < 50%
* Capable of giving informed consent
* Willing and able to comply with the test program as directed by staff.

Exclusion Criteria:

* Subject is not fluent in written or spoken English
* Has physical impairment that prevents the subject from being able to walk or stand
* Is acutely ill/medically complicated, as determined by the investigator.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Recovery Time | 30 minutes
  The time it takes to return to 0 on the Borg Dyspnoea Scale ("No difficulty breathing") following exercise. This is a scale that asks you to rate the difficulty of your breathing. It starts at number 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knuesel, PhD, Principal Investigator — Koronis Biomedical Technologies

IPD SHARING:
Plan to Share IPD: No